CLINICAL TRIAL: NCT01727076
Title: A Phase 1 Study of Recombinant Human IL15 (rhIL15) in Adults With Advanced Solid Tumors: Melanoma, Renal Cell, Non-Small Cell Lung and Squamous Cell Head and Neck Cancer
Brief Title: Recombinant Interleukin-15 in Treating Patients With Advanced Melanoma, Kidney Cancer, Non-small Cell Lung Cancer, or Squamous Cell Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02205; NCI-2012-02205 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CITN11-02; CITN11-02 (Other: Cancer Immunotherapy Trials Network); CITN11-02 (Other: CTEP); U01CA154967 (NIH)
Record Dates: First submitted 2012-11-12; First posted 2012-11-15 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Recurrent Head and Neck Carcinoma; Recurrent Non-Small Cell Lung Carcinoma; Recurrent Renal Cell Carcinoma; Recurrent Skin Carcinoma; Stage III Renal Cell Cancer; Stage IIIA Cutaneous Melanoma AJCC v7; Stage IIIA Non-Small Cell Lung Cancer AJCC v7; Stage IIIB Cutaneous Melanoma AJCC v7; Stage IIIB Non-Small Cell Lung Cancer AJCC v7; Stage IIIC Cutaneous Melanoma AJCC v7; Stage IV Cutaneous Melanoma AJCC v6 and v7; Stage IV Non-Small Cell Lung Cancer AJCC v7; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Melanoma | interventions — Interleukin-15

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (recombinant interleukin-15) (Experimental): Patients receive recombinant interleukin-15 SC daily on days 1-5 of weeks 1 and 2. Treatment repeats every 28 days (4 weeks) for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Biological: Recombinant Human Interleukin-15

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Biological: Recombinant Human Interleukin-15 — Given SC
  Other Names: IL15; Interleukin 15; rhIL-15; rIL15

SUMMARY:
This phase I trial studies the side effects and best dose of recombinant interleukin-15 in treating patients with melanoma, kidney cancer, non-small cell lung cancer, or head and neck cancer that has spread to other places in the body and usually cannot be cured or controlled with treatment. Recombinant interleukin-(IL)15 is a biological product, a protein, made naturally in the body and when made in the laboratory may help stimulate the immune system in different ways and stop tumor cells from growing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of recombinant human IL15 (rhIL15) administered subcutaneously.

SECONDARY OBJECTIVES:

I. To determine the effect of the dose schedules of rhIL15 on the number and phenotype of peripheral blood mononuclear cells including: total white blood cell count; absolute lymphocyte count (ALC); and total number of T cells and natural killer (NK) cells, as well as activated T cells, T cell subsets and NK cell subsets.

II. To determine the effects of the dose schedules of rhIL15 on the function of peripheral blood mononuclear cells including: T cell subset response to recall viral antigens including cytomegalovirus (CMV) and influenza A virus; T cell responses to non-physiologic stimuli including: phytohemagglutinin (PHA); and NK cell cytokine (interferon gamma [IFN-y]) secretion and degranulation by cluster of differentiation 107a (CD107a) expression.

III. To assess tumor response rate by objective response rate (ORR). IV. To assess the immunogenicity, pharmacokinetic (PK) and pharmacodynamic (PD) profiles of National Cancer Institute (NCI) rhIL15.

OUTLINE: This is a dose-escalation study.

Patients receive recombinant interleukin-15 subcutaneously (SC) daily on days 1-5 of weeks 1 and 2. Treatment repeats every 28 days (4 weeks) for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histological or cytological confirmed malignancy in the following disease groups: melanoma, non-small cell lung carcinoma, renal cell carcinoma or squamous cell head and neck carcinoma, for which no standard effective or curative options are available
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Documented evidence of disease progression during 6 month period prior to the time of enrollment
* Prior therapy requirements:

  * At least >= 1 prior completed chemotherapy regimen including chemotherapy, biologic, immunologic or targeted therapy
  * At least 4 weeks from last dose of prior chemotherapy with resolution of the acute toxic effects of the therapy
  * At least 2 weeks from completion of prior radiation therapy
  * At least 4 weeks from last dose of prior investigational therapy
  * Not receiving any current anti-cancer therapy
  * At least 4 weeks from last dose of interferon or IL-2 therapy
  * At least 8 weeks from completion of antibody therapy with anti-checkpoint antibodies, such as anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA4) and anti-programmed cell death 1 (PD1)
  * At least 4 weeks from last dose of prior other biologic agents
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 (Karnofsky > 70%)
* Absolute lymphocytes > 500/mcL
* Absolute neutrophil count > 1,000/mcL
* Platelets > 100,000/mcL
* Total bilirubin within normal institutional limits
* Prothrombin time (PT)/partial thromboplastin time (PTT) < 1.5 x upper limit of normal (ULN)
* Hemoglobin (Hgb) > 9 g/dL
* Alkaline phosphatase =< 2.5 x ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 2 x institutional upper limit of normal
* Serum creatinine < 1.5 x ULN or creatinine clearance > 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* No known central nervous system (CNS) metastases or neurological symptoms possibly related to active CNS metastasis
* Females of childbearing potential must have a negative pregnancy test within 48 hours prior to initiation of protocol therapy; NOTE: subjects are considered not of child bearing potential if they are surgically sterile, they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy or they are postmenopausal; menopause is the age associated with complete cessation of menstrual cycles, menses, and implies the loss of reproductive potential; by a practical definition, it assumes menopause after 1 year without menses with an appropriate clinical profile at the appropriate age; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) from the time the consent is signed and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; women of child-bearing potential and men treated or enrolled on this protocol must also agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) 4 months after completion of rhIL15
* Ability to understand and the willingness to sign a written informed consent document
* No history of any hematopoietic malignancy
* No active (as defined by requiring immunosuppressive therapy) or history of clinically significant autoimmune disease (as defined by previously requiring immunosuppressive therapy)
* No evidence of a clinically significant active infection
* No systemic or inhaled corticosteroids within 7 days prior to initiation of protocol therapy; NOTE: use of topical corticosteroids and/or eye drops containing glucocorticosteroids is acceptable
* No immunosuppressive therapy within 30 days prior to initiation of protocol therapy
* No history of severe asthma, as defined by prior or current use of systemic corticosteroids for disease control, with the exception of physiological replacement doses of cortisone acetate or equivalent, as defined by a dose of 10 mg or less; NOTE: history of mild asthma not requiring daily therapy is eligible
* No history of pulmonary disease such as emphysema or chronic obstructive pulmonary disease (COPD), (forced expiratory volume in one second [FEV1] > 2L or >= 50% of predicted for height and age); pulmonary function tests (PFTs) are required in patients with significant pulmonary or smoking history
* No history of human immunodeficiency virus (HIV), active or chronic hepatitis B, hepatitis C or human T-cell lymphotropic virus (HTLV-I) infection; NOTE: a positive hepatitis B serology indicative of previous immunization (i.e., hepatitis B surface antibody [HBsAb] positive and hepatitis B core antibody [HBcAb] negative), or a fully resolved acute hepatitis B virus (HBV) infection is not an exclusion criterion
* Females of childbearing potential and males must be willing to use an effective method of contraception (hormonal, barrier method of birth control or abstinence) from the time the consent is signed, during the duration of study participation and 4 months after discontinuation of protocol therapy
* Females must not be breastfeeding
* No evidence of clinically significant congestive heart failure, (ejection fraction of 45% or greater)
* No platelet or blood transfusions within two weeks of obtaining baseline laboratory values
* No blood modifiers while enrolled in the study (i.e., growth factors such as erythropoiesis-stimulating agent [ESA] or filgrastim [G-CSF]); NOTE: blood transfusions are allowed per institutional guidelines

Exclusion Criteria:

* Patients who have had chemotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C), or radiotherapy within 2 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Class II or greater congestive heart failure as described in the New York Heart Association Functional Classification criteria
* Patients with thyroid disease should be excluded unless their T4 is normal or they are on replacement therapy
* Patients with primary brain cancer or known brain metastases should be excluded from this clinical trial
* Patients who have received prior anti-CTLA4 or anti-PD1 therapy less than 8 weeks prior to enrollment
* Patients who have received prior biologic agents less than 4 weeks prior to enrollment
* Patients who have received prior interferon or IL-2 therapy less than 4 weeks prior to enrollment
* ECOG score greater than 1 (Karnofsky < 70%)
* HIV-positive patients
* Positive hepatitis C serology
* Patients who are receiving any other investigational agents
* Inability to home monitor blood pressure
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02-15 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
MTD defined as the next lower dose in which 1 or more patients experiences a dose limiting toxicity defined as grade 3 or 4 toxicity graded according to the NCI Common Terminology Criteria for Adverse Events version 4.0 | 28 days

SECONDARY OUTCOMES:
ALC, monitored daily during treatment | Up to 6 months
  The absolute increase in each cell subset as well as the variance in change across each dose level (mean, median, and SE/SD will be reported for each dose level and ALC, circulating NK count, and circulating CD4/CD8 cell counts).
Change in NK cell function measured using flow cytometric analysis of cytokine (IFN-y) secretion and expression of degranulation marker CD107a | Baseline to day 15
  The absolute change in responses for each patient will be calculated by subtracting the SFC/million PBMC at day 11 from the SFC/million PBMC at baseline for each antigen.
Change in presence of auto-antibodies, assessed by ELISA | Baseline to day 4 of week 2
  The number and percentage of patients developing auto-antibodies to IL15 will be tabulated by dose cohort.
Change in T cell responses to non- physiologic stimuli including PMA | Baseline to day 4 of week 2
  The absolute change in responses for each patient will be calculated by subtracting the SFC/million PBMC at day 11 from the SFC/million PBMC at baseline for each antigen.
Change in T cell subset response to recall viral antigens including CMV and influenza A virus, determined by enzyme-linked immunosorbent spot assay | Baseline to day 4 of week 2
  The absolute change in responses for each patient will be calculated by subtracting the spot forming cells (SFC)/million peripheral blood mononuclear cell (PBMC) at day 11 from the SFC/million PBMC at baseline for each antigen.
Change in total number of T cells and NK cells, as well as activated T cells, T cell subsets, and NK cell subsets, assessed by flow cytometric analysis of peripheral blood mononuclear cells | Baseline to day 15
  The percentage of cells positive for the marker and/or mean fluorescence intensity (MFI) at time points after rhIL15 administration will be compared to baseline and the change will be calculated as %after/ %baseline or MFI after/ MFI baseline.
ORR based on RECIST criteria | Up to day 56 (after 2 courses)
  Percentages and exact 2-sided 95% confidence intervals of the numbers in each of the overall response categories (complete response, partial response, stable disease and progressive disease) will be calculated for each dose cohort.
Serum PK of IL15 and IL15 receptor-alpha, assessed by enzyme linked immunosorbent assay (ELISA) | Pre-dose, and 10 minutes, 1, 4, and 24 hours after administration
  IL15 and IL15 receptor-alpha levels will be plotted over time for each dose group.
Total white blood cell count, monitored daily during treatment | Up to 6 months
  The absolute increase in each cell subset as well as the variance in change across each dose level (mean, median, and standard error [SE]/standard deviation [SD] will be reported for each dose level and absolute lymphocyte count [ALC], circulating NK count, and circulating CD4/CD8 cell counts).

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Miller, Principal Investigator — Cancer Immunotherapy Trials Network
Locations (5):
- United States (5):
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

REFERENCES:
- [Derived] Margolin K, Morishima C, Velcheti V, Miller JS, Lee SM, Silk AW, Holtan SG, Lacroix AM, Fling SP, Kaiser JC, Egan JO, Jones M, Rhode PR, Rock AD, Cheever MA, Wong HC, Ernstoff MS. Phase I Trial of ALT-803, A Novel Recombinant IL15 Complex, in Patients with Advanced Solid Tumors. Clin Cancer Res. 2018 Nov 15;24(22):5552-5561. doi: 10.1158/1078-0432.CCR-18-0945. Epub 2018 Jul 25. PMID 30045932
- [Derived] Miller JS, Morishima C, McNeel DG, Patel MR, Kohrt HEK, Thompson JA, Sondel PM, Wakelee HA, Disis ML, Kaiser JC, Cheever MA, Streicher H, Creekmore SP, Waldmann TA, Conlon KC. A First-in-Human Phase I Study of Subcutaneous Outpatient Recombinant Human IL15 (rhIL15) in Adults with Advanced Solid Tumors. Clin Cancer Res. 2018 Apr 1;24(7):1525-1535. doi: 10.1158/1078-0432.CCR-17-2451. Epub 2017 Dec 4. PMID 29203590